CLINICAL TRIAL: NCT03688945
Title: Art Heals - (the Effects of Art After Robot Assisted Surgery)
Brief Title: Art in Improving Outcomes in Participants Undergo Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Art gallery dissembled- no research goals with new art.
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 43217; NCI-2018-00457 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 43217 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-09-19; First posted 2018-09-28 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Health Status Unknown
MeSH Terms: interventions — Art Therapy; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (art sessions) (Experimental): Participants attend at least 1 session of viewing art pieces over 15 minutes every day for 2 years.
  Interventions: Procedure: Art Therapy; Other: Questionnaire Administration
- Arm II (standard of care) (Active Comparator): Participants receive standard of care for 2 years.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Art Therapy — Attend art viewing sessions
  Arms: Arm I (art sessions)
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm II (standard of care)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well art works in improving outcomes in participants who are undergoing surgery. Exposure to art may help to improve clinical and psychological outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Investigate through evidence-based randomized controlled trial the effect of exposure to art during the perioperative period on the outcome of surgical outcomes II. Assess patient response to artwork and investigate the correlation of patient response with the clinical outcomes of the patients.

III. Measure cognitive changes that may occur for patients based on art exposure.

OUTLINE: Participants are randomized into 1 of 2 arms.

ARM I: Participants attend at least 2 sessions of viewing art pieces over 15 minutes every day for 2 years.

ARM II: Participants receive standard of care for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant inpatients that will stay for at least 2 days postoperatively and do not require continuous monitoring
* All races and ethnic groups are eligible for this study

Exclusion Criteria:

* Patients with altered mental status, psychiatric illness, debilitating pain, blind patients, or those who require continuous monitoring postoperatively will be excluded from the study
* Adult unable to consent, individuals who are not yet adults, pregnant women or prisoners

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Mental health wellbeing score | Up to 2 years
  Will be assessed by using a Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS). This is a 14 item scale with 5 response categories that cover both feeling and functioning aspects of mental wellbeing.

SECONDARY OUTCOMES:
Reduced pain: NRS | Up to 2 years
  Will assess by using a validated visual numeric rating scale - corresponding to pain experienced over 24 hours
Anxiety score (patient) | Up to 2 years
  Will be assessed by using State Trait Inventory for Adults (STAI). - A self reporting survey which measures anxiety.
Hope score | Up to 2 years
  Will be assessed by using Herth Hope Index. A 12 item self reporting questionnaire measuring the sense of hope.
Change in blood pressure | Up to 2 years
  Will assess systolic and diastolic pressure . Parameters will be collected from the patient chart
change in recovery of bowel function | Up to 2 years
  Evaluated using Parameters collected from the patient chart

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid Guru, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States